CLINICAL TRIAL: NCT06337682
Title: Describing the Management of Hypertension in a UK Care Home Population
Brief Title: Blood Pressure Management in the Care Home Population
Acronym: BPITCH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Oliver Todd, Academic Clinical Lecturer, University of Leeds
Other Study IDs: CB_CY_P09_23_11
Record Dates: First submitted 2024-03-14; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Aging; Hypertension
Keywords: Nursing Home; Residential Home; Deprescribing
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Care home cohort: Individuals aged 65 or over registered to a GP practice which is part of the Connected Bradford Database who have been admitted to a CH between January 2016 and January 2020, with a recorded length of stay more than 6 weeks, will be included in the study.

SUMMARY:
The UK care home population is projected to increase significantly over the coming decades. A high proportion of individuals in a care home have multiple long-term conditions and take large amounts of prescribed medication. This means they are routinely excluded from research studies and so there is little evidence on which to base treatment of long-term conditions such as high blood pressure. Furthermore, given that 1 in 4 people admitted into a care home die within 1 year, the benefit of treating high blood pressure to reduce the risk of heart attack or stroke must be balanced with the need to optimise quality of life. The aim of this study is to describe the health and social characteristics of the UK care home population with a particular focus on the management of blood pressure in the population. It is hoped that the findings of this study will help inform future research into the management of chronic conditions in care home residents.

DETAILED DESCRIPTION:
The investigators will use the connected Bradford dataset to examine UK electronic health records to describe the UK care home population and management of hypertension in this population. The sample will include all adults aged 65 and over who have been admitted into a care home between January 2016 and December 2019. The investigators will extract data at the time of care home admission including age, sex, ethnicity, coded diagnosis of hypertension, indices of frailty and risk of falls as well as comorbidities relevant to cardiovascular risk and falls risk. Analysis will include looking at the prevalence of hypertension amongst the care home population, describing treatment patterns (i.e. number and type of prescribed anti-hypertensive medications, frequency of blood pressure monitoring) and the proportion of patients with blood pressure controlled according to National Institute of Health and Care Excellence (NICE) guidelines. The investigators will also look to establish whether there are any changes in the number and type of prescribed antihypertensive medication before and after admission to a care home (i.e. intensification of pharmacological therapy or deprescribing) and whether this differs amongst different subgroups of populations including patients with terminal illness and stroke diagnosis. The investigators will also estimate frequency of falls in the year following care home admission.

ELIGIBILITY:
Inclusion Criteria:

* registered to a GP practice contributing to the Connected Bradford dataset at the point of admission
* a recorded length of stay in a care home of longer than six weeks
* recorded social care entry for nursing or residential care in the Bradford council social care data.

Exclusion Criteria:

* no exclusion criteria applied to keep the sample representative of the real-world care home population.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Care home residents in the Bradford metropolitan area. The Bradford population has high levels of deprivation and ethnic diversity; a large proportion of the population identify as Pakistani ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of blood pressure measurements | from the point of admission up to 12 months following admission
  the proportion of individuals entering a care home, with a diagnosis of hypertension, have their blood pressure measured in the year following admission
change in antihypertensive medication | 6 months before admission to 6 months following admission
  change in the number or type of antihypertensive mediation from six months before care home admission to six months following care home admission
Injurious falls | from the point of admission up to 12 months after admission
  one year incidence of a fall resulting in hospital attendance in those entering a care home

SECONDARY OUTCOMES:
Prevalence of hypertension | at the day of admission to a care home (this will vary between each individual)
  the proportion of individuals in the care home cohort with a diagnosis of hypertension at the point of care home admission
Antihypertensive medication | at the day of admission to a care home (this will vary between each individual)
  the number and type of antihypertensive medication prescribed at the point of admission
Blood pressure treatment | 12 months following admission
  of those with a diagnosis of hypertension and a blood pressure value recorded in the 12 months after admission, proportion a blood pressure value below the target set by the National Institute for Health and Care Excellence (i.e. for those aged 80 and over 150/90 and those aged below 80 years 140/90)

OTHER OUTCOMES:
change in systolic pressure following care home admission | 12 months before admission for the first measure and 12 months after admission for the second measure.
  the difference between systolic blood pressure recorded before care home admission (defined as less than 12 months for care home admission) and systolic blood pressure recorded after care home admission (blood pressure recorded within 12 months following admission)

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Unit for Ageing and Stroke Research, Bradford, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
using anonymised routine health data so cannot be shared. Will share code used to identify cohort with identifiers removed